CLINICAL TRIAL: NCT04693793
Title: Establishing Clinical Utility for a New Diagnostic Test for Patients With Shortness of Breath: A CPV® Randomized Controlled Trial
Brief Title: Establishing Clinical Utility for a New Diagnostic Test for Patients With Shortness of Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-ACT-2020
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Dyspnea; Unexplained Chronic Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: The study will enroll specialist physicians, specifically cardiologists and pulmonologists, practicing in the US. Participants are randomly assigned to either a control, intervention 1, or intervenion 2 arm upon enrollment. All eligible and consented participants will complete two rounds of three patient simulations.
  The intervention 1 and intervention 2 arms only will receive educational material about the Janssen test in between these two rounds. Intervention 1 arm participants only will receive the Janssen test results whether they select it or not, and Intervention 2 participants will receive the Janssen test results only if they select it in the second round of simulated cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): These providers will complete two rounds of three simulated patient cases (CPVs). Control arm physicians will continue to have access to standard of care diagnostic tools, but not the Janssen test results.
- Educational Materials and Janssen Test Results (Intervention 1) (Experimental): Participants will care for the same set of CPV patients as the control arm, but will be educated on and will receive the Janssen test results whether they select it or not. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Other: Education Materials and Janssen Test
- Educational Materials and Janssen Test Results when Selected (Intervention 2) (Experimental): Participants will care for the same set of CPV patients as the control arm, but will be educated on and will receive the Janssen test results only if they select it. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Other: Education Materials and Janssen Test

INTERVENTIONS:
Other: Education Materials and Janssen Test — Intervention-1- and Intervention-2-arm participants will receive educational materials duplicating what physicians would receive in the real-world market as they adopt the Janssen technology. These materials are comprised of a slide deck, a sample test report, and a frequently asked questions (FAQ) sheet.
  Intervention 1 participants only will receive the Janssen test results whether they select it or not, and Intervention 2 participants will receive the Janssen test results only if they select it during the second round of case simulations.
  Arms: Educational Materials and Janssen Test Results (Intervention 1); Educational Materials and Janssen Test Results when Selected (Intervention 2)

SUMMARY:
This study will collect high-quality data on how practicing specialist physicians, specifically cardiologists and pulmonologists, across the U.S. currently manage patients with unexplained chronic dyspnea and and how the results of Janssen Pharmaceuticals' test change clinical decision making. To do so, this study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions.

DETAILED DESCRIPTION:
This study will collect high-quality data on how practicing specialist physicians, specifically cardiologists and pulmonologists, across the U.S. currently manage patients with unexplained chronic dyspnea and and how the results of Janssen Pharmaceuticals' test change clinical decision making. Data from this study will better illuminate the clinical use cases in which the Janssen test has the most significant impact on clinical decision making (and thus the largest potential clinical utility) and the associated physician characteristics (e.g., age, practice setting, training) associated with test adoption.

This study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions. CPVs are a unique and scalable tool that standardizes practice measurement by having all providers care for the same (virtual) patients. With all providers caring for the same patients, the CPVs generate unbiased data that yields powerful insights into clinical decision making and how these decisions change with the introduction of a new product or solution. Data from the CPVs can quickly demonstrate the clinical utility of a solution, be published in peer-reviewed literature, inform marketing strategies and positively impact coverage and reimbursement decisions.

The study is a prospective cohort trial with six steps:

1. Enrollment: The study will enroll 249 cardiologists and pulmonologists practicing in the U.S. who are determined to be eligible by an eligibility screener.
2. Provider survey: Once the participants are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background.
3. Randomization: The 249 participants will be randomized into three equally-sized arms (83 participants each arm): Control, Intervention 1, and Intervention 2.
4. CPVs (First Round): Participants will complete three randomly-assigned CPV patient simulations. Cases will be identical across the intervention and control arms. All interactive cases are presented on an online platform, and are accessible via unique weblinks and any internet-connected computer.
5. Education: The Intervention-1- and Intervention-2-arm participants will receive educational materials duplicating what physicians would receive in the real-world market as they adopt the Janssen technology. These materials are comprised of a slide deck, a sample test report, and a frequently asked questions (FAQ) sheet.
6. CPVs (Second Round): All participating physicians will then be asked to complete three additional CPV patient simulations. The cases are given to the doctors in a random order. Cases will be identical across the intervention and control arms. At an appropriate point in each case, Intervention 1 participants only will receive the Janssen test results whether they select it or not, and Intervention 2 participants will receive the Janssen test results only if they select it. Control arm participants will continue to have access to standard of care diagnostic tools, but not the Janssen test. All cases are presented on an online platform, and participants are provided with unique weblinks, accessible via any internet-connected computer.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified cardiologist or pulmonologist for at least two years
2. Averaging at least 20 hours per week of clinical and patient care duties over the last six months
3. Routinely evaluate patients for unexplained or chronic dyspnea in their practice
4. Practicing in the U.S.
5. English speaking
6. Access to the internet
7. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Practicing in an academic setting
3. Unable to access the internet
4. Not practicing in the U.S.
5. Not averaging at least 20 hours per week of clinical or patient care duties over the last six months
6. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
CPV-measured clinical score difference | 3 months
  Difference-in-differences regression analysis between the control and the intervention groups' diagnosis and treatment of chronic dyspnea, as measured by the participants diagnostic and treatment CPV case domain scores. In each domain of a CPV (history, physical exam, workup, diagnosis and treatment), participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum from 0 to a high potential score of up to 100 percent in each domain, where higher scores mean better outcomes.
Test Adoption Rate | 3 months
  Rate of adoption of the Janssen test in Intervention 2 arm participants.
CPV-measured cost difference | 3 months
  Difference in expected cost of care between control and intervention participants. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs.)

SECONDARY OUTCOMES:
CPV-measured clinical score differences by use case | 3 months
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention participants. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is a average score of the subcategory scores (percent correct). This will be examined for each of the use cases to determine in which case(s) CPV scores most improved.
CPV-measured cost differences by use case | 3 months
  Difference in expected cost of care between control and intervention participants. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs.) This will be examined for each of the use cases to determine in which case(s) cost metrics most improved.
CPV-measured baseline variation | 3 months
  Participants completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD PhD, Principal Investigator — President, QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Result] Burgon TB, Cox-Chapman J, Czarnecki C, Kropp R, Guerriere R, Paculdo D, Peabody JW. Engaging Primary Care Providers to Reduce Unwanted Clinical Variation and Support ACO Cost and Quality Goals: A Unique Provider-Payer Collaboration. Popul Health Manag. 2019 Aug;22(4):321-329. doi: 10.1089/pop.2018.0111. Epub 2018 Oct 17. PMID 30328782
- [Result] Peabody JW, Strand V, Shimkhada R, Lee R, Chernoff D. Impact of rheumatoid arthritis disease activity test on clinical practice. PLoS One. 2013 May 7;8(5):e63215. doi: 10.1371/journal.pone.0063215. Print 2013. PMID 23667587
- [Result] Peabody J, Martin M, DeMaria L, Florentino J, Paculdo D, Paul M, Vanzo R, Wassman ER, Burgon T. Clinical Utility of a Comprehensive, Whole Genome CMA Testing Platform in Pediatrics: A Prospective Randomized Controlled Trial of Simulated Patients in Physician Practices. PLoS One. 2016 Dec 30;11(12):e0169064. doi: 10.1371/journal.pone.0169064. eCollection 2016. PMID 28036350
- [Result] Solon O, Woo K, Quimbo SA, Shimkhada R, Florentino J, Peabody JW. A novel method for measuring health care system performance: experience from QIDS in the Philippines. Health Policy Plan. 2009 May;24(3):167-74. doi: 10.1093/heapol/czp003. Epub 2009 Feb 18. PMID 19224955
- [Derived] de Belen E, McConnell JW, Elwing JM, Paculdo D, Cabaluna I, Linder J, Peabody JW. Gaps in the Care of Pulmonary Hypertension: A Cross-Sectional Patient Simulation Study Among Practicing Cardiologists and Pulmonologists. J Am Heart Assoc. 2023 Jan 17;12(2):e026413. doi: 10.1161/JAHA.122.026413. Epub 2023 Jan 11. PMID 36628980